CLINICAL TRIAL: NCT00588094
Title: A Phase II Study of Dose Augmented Rituximab and Ice for Patients With Primary Refractory and Poor Risk Relapsed Aggressive B-Cell Non-Hodgkin's Lymphoma Undergoing Second-Line Therapy Prior to Stem Cell Transplantation
Brief Title: Dose Augmented Rituximab and ICE for Pts With Primary Refractory and Poor Risk Relapsed Aggressive B-Cell NHL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-075
Record Dates: First submitted 2007-12-26; First posted 2008-01-08 (Estimated); Results first posted 2015-12-04 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-10

CONDITIONS: Lymphoma; B-cell Non-Hodgkin's Lymphoma
Keywords: Lymphoma; ASCT; B-cell non-Hodgkin's lymphoma; Cancer; Second line therapy; ICE; Stem cell transplant
MeSH Terms: conditions — Lymphoma; Lymphoma, B-Cell; Neoplasms | interventions — Rituximab; Ifosfamide; Carboplatin; Etoposide; Mesna; Granulocyte Colony-Stimulating Factor; Stem Cell Transplantation; Filgrastim; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): R-ICEesc will be administered with the intent of administering 2 cycles, each 21 days apart admixed with 4 doses of rituximab. G-CSF will be administered at 960 ug or 10 ug/kg if patient is > 100 kg after cycles one and two for PBPC collection for the first 10 patients enrolled. G-CSF will be administered in standard dosing for cycle one and then at 960 ug or 10 ug/kg (if patient is > 100 kg) after cycle two for PBPC collection for the remaining 22 patients. All responding patients who make at least 2 x 106 CD34+ cells/kg will receive high dose therapy and ASCT on other protocols.
  Interventions: Drug: Rituximab, Ifosfamide, Carboplatin, VP-16, Mesna, G-CSF, Stem Cell Transplant

INTERVENTIONS:
Drug: Rituximab, Ifosfamide, Carboplatin, VP-16, Mesna, G-CSF, Stem Cell Transplant — ANC must be ≥1000/µl and platelet count must be ≥50,000/µl. Rituximab will be administered at a dose of 375 mg/m2 IV on days 1 and 3 of the each cycle. Premedication will be given.ICE will be administered as follows: Day 3: Etoposide 200 mg/m2 IV q12 hrs x 3. Day 4: Ifosfamide 10 g/m2 and MESNA 10 g/m2 mixed and infused together as a continuous infusion over 48 hours. Day 5: Carboplatin IV dosed by the Calvert formula using an AUC of 5.
  Carboplatin dose (mg) = 5 x (Clcr + 25) For the first ten patients enrolled, G CSF will be administered beginning on day seven of each cycle and G CSF will continue until stem cell collection is completed. The dose will be 960 ug or 10 ug/kg if weight is greater than 100 kg.
  For the remaining patients, G-CSF will be administered for 10 days beginning on day 7 for cycle 1. The dose will be 300-480 ug/d. For cycle 2 the dose will be 960 ug or 10ug/kg if weight is > 100kg. Leukapheresis will continue.
  Other Names: ASCT,Rituxan, Ifex, Paraplatin®, etoposide, Vepesid®, Mesnex®, Neupogen, Neulasta

SUMMARY:
The purpose of this research is to study a treatment program for patients with aggressive lymphoma that has come back after initial or first therapy (called relapsed) or that has not responded to first therapy (called refractory). Since 1993, we have used a combination of chemotherapy known as ICE (Ifosfamide, Carboplatin, and Etoposide) for your type of lymphoma. In many patients, this treatment helps the disease to shrink before giving high-dose therapy and autologous stem cell transplant (ASCT). Only patients who respond to these types of treatments have a chance of their disease going away (remission) with an ASCT. In 1999, we studied the same treatment but added another medicine for your type of lymphoma, Rituximab (Rituxan), to the ICE treatment (RICE). More patients had lymphoma shrinkage from this treatment (chemosensitive disease) than with ICE alone. These patients then received high dose therapy and autologous stem cell transplant and have an improved chance of having a remission.

ICE chemotherapy is standard chemotherapy used at Memorial Sloan-Kettering Cancer Center. However, it is different in this study because of the higher doses. We are testing higher doses of RICE treatment for patients in this study.

In our current study in Hodgkin's lymphoma, we are giving these higher doses of ICE (called augmented ICE) to patients who also have higher risk. We hope to show in this study that by using Rituximab and augmented ICE that we can improve your ability to achieve a remission (that is, to have the disease go away).

DETAILED DESCRIPTION:
The purpose of this study is to determine if dose escalation of the rituximab-ICE (RICEesc) program can improve the overall response rate of patients with primary refractory or poor risk relapsed aggressive B cell lymphoma. R-ICEesc will be administered for 2 cycles with peripheral blood progenitor cells (PBPCs) collected after cycle 2.

A two-stage design will be employed, such that the study will be terminated if in the first cohort of patients it appears that the overall response rate is <50% or if >25% patients fail to mobilize at least 2 x 106 CD34+ cells/kg.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of the one of the following B cell aggressive lymphomas, confirmed by an MSKCC pathologist: Diffuse Large, Immunoblastic, Mantle cell, Anaplastic Large Cell, De novo transformation of follicular lymphoma, or classical Hodgkin's lymphoma which is CD20 antigen positive.
* Tumors must stain positive for CD20.
* Primary refractory disease proven by biopsy or fine needle aspiration (cytology) of an involved site
* Relapsed diffuse large, immunoblastic, anaplastic, de novo transformation of follicular lymphoma, or classical Hodgkin's lymphoma which is CD20 antigen positive proven by biopsy or fine needle aspiration (cytology) of an involved field site and at least two of the three following risk factors: LDH> upper limit of normal, KPS < 80%, Stage III or IV disease.
* All mantle cell lymphoma patients in first relapse
* Failure of doxorubicin or mitoxantrone containing front-line therapy
* Bidimensionally measurable disease.
* Cardiac ejection fraction of greater than 50%, measured since last chemotherapy.
* Serum creatinine <1.5 mg/dl; if creatinine >1.5 mg/dl then the measured 12- or 24-hour creatinine clearance must be >60 ml/minute.
* ANC>1000/µl and Platelets>50,000/µl
* Total bilirubin < 2.0 mg/dl in the absence of a history of Gilbert's disease.
* Females of childbearing age must be on an acceptable form of birth control.
* Age between 18 and 72
* HIV I and II negative.
* Patients or their guardians must be capable of providing informed consent.

Exclusion Criteria:

* Any lymphoma subtype other than those described among the inclusion criteria.
* All patients with relapsed diffuse large, immunoblastic, anaplastic, de novo transformation of follicular lymphoma, or classical Hodgkin's lymphoma which is CD20 antigen positive disease who have <2 of following risk factors: LDH> upper limit of normal, KPS < 80%, Stage III or IV disease.
* History of second-line chemotherapy
* Presence of CNS involvement.
* Prior treatment with carboplatin, cisplatin, ifosfamide, or etoposide
* Hepatitis B surface antigen positive.
* Known pregnancy or breast-feeding.
* Medical illness unrelated to NHL, which in the opinion of the attending physician and/or principal investigator will preclude administering chemotherapy safely.
* History of any malignancy for which the disease-free interval is <5 years, excluding curatively treated cutaneous basal cell or squamous cell carcinoma and carcinoma in-situ of the cervix

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Moskowitz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering web site — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- R-ICEesc: R-ICEesc will be administered with the intent of administering 2 cycles, each 21 days apart admixed with 4 doses of rituximab. G-CSF will be administered at 960 ug or 10 ug/kg if patient is > 100 kg after cycles one and two for PBPC collection for the first 10 patients enrolled. G-CSF will be administered in standard dosing for cycle one and then at 960 ug or 10 ug/kg (if patient is > 100 kg) after cycle two for PBPC collection for the remaining 22 patients. All responding patients who make at least 2 x 106 CD34+ cells/kg will receive high dose therapy and ASCT on other protocols.
Period: Overall Study
Arm/Group | R-ICEesc
Started | 20
Completed | 15
Not Completed | 5
Not completed — Adverse Event | 3
Not completed — Progression of Disease | 2

BASELINE CHARACTERISTICS:
Arm/Group | R-ICEesc
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Improve the Overall Response Rate
Description: assessing the response rate (CR+PR)
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | R-ICEesc
Number analyzed (Participants) | 17
participants
  Complete Remission | 4
  Complete Remission/Unconfirmed | 2
  Partial Remission | 7
  Progression of Disease | 4

ADVERSE EVENTS:
Arm/Group | R-ICEesc
Serious Adverse Events (participants affected / at risk) | 12/20
Other Adverse Events (participants affected / at risk) | 12/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R-ICEesc (N=20)
Cardiac disorder (Cardiac disorders) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2)
Creatinine increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Delusions (Psychiatric disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 6 (8)
Fever (General disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Infection NOS (Infections and infestations) | 2 (2)
Infection with grade 3/4 neut (Infections and infestations) | 2 (2)
White blood cell decreased (Investigations) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R-ICEesc (N=20)
Blood bilirubin increased (Investigations) | 3 (8)
CPK increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (12)
Anemia (Blood and lymphatic system disorders) | 12 (259)
Hyperglycemia (Metabolism and nutrition disorders) | 11 (51)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (17)
Hypocalcemia (Metabolism and nutrition disorders) | 9 (67)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 7 (11)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (5)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 9 (60)
White blood cell decreased (Investigations) | 12 (136)
Lymphocyte count decreased (Investigations) | 12 (229)
Neutrophil count decreased (Investigations) | 11 (48)
Activated partial thromboplastin time prolonged (Investigations) | 4 (6)
Platelet count decreased (Investigations) | 11 (182)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 3 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes